CLINICAL TRIAL: NCT06256718
Title: Implementation of Evidence-Based Strategies to Optimize HPV Vaccination in Rural Primary Care Settings
Brief Title: Implementation of Evidence-Based Strategy (PC TEACH) for the Optimization of HPV Vaccination in Rural Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I 1998021; NCI-2021-12381 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 1998021 (Other: Roswell Park Cancer Institute); R01MD016850 (NIH)
Record Dates: First submitted 2024-02-02; First posted 2024-02-13 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health services research (PC TEACH) (Other): Primary practice providers sites receive PC TEACH over 3.5 hours for 12 months
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Evidence-based strategy (PC TEACH)
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational

SUMMARY:
This study evaluates the implementation of evidence based strategies to optimize HPV vaccination in rural primary care settings. Some of the largest disparities in human papillomavirus vaccination (HPVV) rates exist in rural communities, which represent missed opportunities for cancer prevention. Primary care provider visits in these communities serve as a crucial opportunity to communicate the importance of timely vaccination that is essential to effective cancer prevention. This study implements and tests a practice-level intervention (PC TEACH) using practice facilitation of evidence-based strategies to expand reach to rural community-based primary care settings to optimize delivery and increase HPVV rates. PC TEACH program may help rural communities overcome access and awareness factors that keep them from receiving HPVV.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify practices from across 20 rural counties in central and western New York (CWNY) using registry data from New York State Immunization Information System.

II. Leverage established community network contacts of primary care practices across 20 rural counties in CWNY to support and enhance recruitment and retention activities.

III. Establish a Rural Cancer Health Equity Community Advisory Board (CAB) to enhance capacity to implement evidence-based cancer prevention activities in rural primary care settings (like primary care practice-level, medical office-based intervention [PC-TEACH] for Human Papilloma Virus Vaccine [HPVV]).

IV. Recruit rural primary care practices to implement PC TEACH intervention and contribute practice, provider, and patient-level data including adolescent vaccination rates.

V. Implement systematic practice-level changes (i.e., PC TEACH strategies) in rural community-based primary care practices.

V. Evaluate effectiveness of PC TEACH intervention and quality improvement within the practices using process and outcome evaluation measures.

OUTLINE:

Primary practice providers sites receive PC TEACH over 3.5 hours for 12 months.

After completion of study, primary care provider sites are followed up for 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* PRACTICES: Are located in the 20-county target region
* PRACTICES: Have an adolescent patient population >= 150 (aged 9-18)
* PRACTICES: Administer adolescent vaccines (e.g., HPV, Tdap, MCV4)
* PRACTICES: Are willing to share aggregate practice and patient-level data (e.g., electronic health record [EHR], surveys)
* PARTICIPANTS: Medical providers and medical staff >= 18 years of age
* PARTICIPANTS: Primary care providers and medical office staff who deliver adolescent care at community-based primary care practice sites across 20 rural counties in central and western New York
* PARTICIPANTS: Age >= 18 years of age (no upper limit)
* PARTICIPANTS: English speaking
* PARENT/GUARDIAN SURVEY: Adult accompanying a child or children aged 9 to 17
* PARENT/GUARDIAN SURVEY: English speaking
* PARENT/GUARDIAN SURVEY: Presenting to the participating clinic for an outpatient well child visit or regular checkup
* PARENT/GUARDIAN SURVEY: Willing to complete an anonymous survey while visiting the clinic

Exclusion Criteria:

* Unwilling or unable to follow protocol requirements
* Adults unable to complete study measures in English
* Individuals who are not yet adults (infants, children, teenagers)
* Cognitively impaired adults/adults with impaired decision-making capacity
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Adolescent HPV vaccination rates | Up to 5 years (60 months)
  To evaluate the impact (short and long-term) of the proposed PC TEACH (primary care practice-level, medical office-based intervention) intervention on human papilloma virus vaccine (HPVV) uptake and completion rates using a staggered (stepped-wedge) intervention schedule. Briefly, practice-specific vaccine rates data will be modeled as a function of time in intervention (0, 6, 12, 18, or 24 months), while adjusting for baseline rates collected prior to intervention for each practice. For vaccine rates, an additional factor for calendar time will be included in the model to address potential seasonal effects.

SECONDARY OUTCOMES:
Age at vaccination | Up to 5 years (60 months)
  will evaluate the impact of the proposed PC TEACH intervention on age at using a staggered (stepped-wedge) intervention schedule. Briefly, practice-specific vaccine rates data will be modeled as a function of time in intervention (0, 6, 12, 18, or 24 months), while adjusting for baseline rates collected prior to intervention for each practice.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Rodriguez, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States